CLINICAL TRIAL: NCT06845670
Title: Effects of Wurn Technique on Symptoms of Dyspareunia, Menstrual Cramps and Quality of Life in Women With Infertility
Brief Title: Effects of Wurn Technique on Dyspareunia, Menstrual Cramps & QoL in Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maha Ashfaq
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Wurn technique
  Interventions: Other: Wurn technique
- Controlled group (Experimental): Pelvic floor relaxation
  Interventions: Other: Wurn technique

INTERVENTIONS:
Other: Wurn technique — Wurn technique is a massage technique and PF relaxation exercises are to relax tighten pelvic floor muscles.
  Other Names: Pelvic floor relaxation exercise

SUMMARY:
Wurn technique is a PT technique. It is site specific massage therapy in the form of relaxing technique, helps to promote the function of abdominopelvic and reproductive organs.

DETAILED DESCRIPTION:
This study will be randomized controlled trial, will be completed in 10 months duration. Non probability Conveninence sampling technique will be used with 54 participants after randomization. Effect will be obseved in 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Women with infertility between age 25 to 45
* women who were unable to conceive for 12months with regular unprotected intercourse
* women with infertility indicating sexual pain, irregular periods with menstrual cramps.
* women with secondary infertility

Exclusion Criteria:

* Women with active infections and abnormal ovarian cysts.
* Any abdominopelvic surgery within last 90days.
* Any medical history of active abdominopelvic cancer or malignancy.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 54 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index Scoring | 2weeks duration
  Measure sexual functioning of women in six domains: desire, arousal, lubrication, orgasm, satisfaction and pain
Mankoski Pain Scale | 2weeks duration
  Numerical pain scale ranging from 0 to 10
FertiQoL | 2weeks duration
  Asses quality of life of an individual with infertility

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No